CLINICAL TRIAL: NCT00410488
Title: Dose/Schedule Finding Study of Palonosetron in Sarcoma Patients Receiving Multi-Day Chemotherapy With Adriamycin and Ifosfamide (AI)
Brief Title: Palonosetron in Sarcoma Patients Receiving Chemotherapy With Adriamycin and Ifosfamide (AI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005-0664
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-02

CONDITIONS: Sarcoma; Nausea; Vomiting
Keywords: Sarcoma; Palonosetron; Aloxi; Nausea; Vomiting
MeSH Terms: conditions — Sarcoma; Nausea; Vomiting | interventions — Palonosetron; Doxorubicin; Ifosfamide; Dexrazoxane; Mesna; Vincristine; Dexamethasone; Calcium Dobesilate; dexamethasone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palonosetron - 1 Dose (Active Comparator): Arm 1: Palonosetron 0.25 mg intravenous (IV) for 1 dose (day 0).
  Dexamethasone: IV piggyback daily for 5 days (12 mg on day 0, and 8 mg on days 1-4) 30 minutes prior to chemotherapy. Chemotherapy treatment regimen: Zinecard: 750 mg/m2 as an IV bolus; Doxorubicin: 75 mg/m2 as an IV bolus OR 75 mg/m2 as continuous IV infusion over 72 hours (without zinecard) on Day 0. Mesna: 500 mg/m2 given simultaneously with ifosfamide day 0; then 1500 mg/m2 over 24 hours for days 0, 1, 2, and 3 (infusion completing on day 4); Ifosfamide: 2.5 g/m2 IV bolus over 3 hours; days 0, 1, 2, 3 (total dose = 10 g/m2); Vincristine: 2 mg IV by rapid administration on day 0 (for patients with small cell histology).
  Interventions: Drug: Palonosetron - Single Dose; Drug: Adriamycin; Drug: Ifosfamide chemotherapy (AI); Drug: Zinecard; Drug: Mesna; Drug: Vincristine; Drug: Dexamethasone
- Palonosetron - 3 Doses (Active Comparator): Arm 2: Palonosetron 0.25 mg IV for 3 doses (days 0, 2, 4).
  Dexamethasone: IV piggyback daily for 5 days (12 mg on day 0, and 8 mg on days 1-4) 30 minutes prior to chemotherapy. Chemotherapy treatment regimen: Zinecard: 750 mg/m2 as an IV bolus; Doxorubicin: 75 mg/m2 as an IV bolus OR 75 mg/m2 as continuous IV infusion over 72 hours (without zinecard) on Day 0. Mesna: 500 mg/m2 given simultaneously with ifosfamide day 0; then 1500 mg/m2 over 24 hours for days 0, 1, 2, and 3 (infusion completing on day 4); Ifosfamide: 2.5 g/m2 IV bolus over 3 hours; days 0, 1, 2, 3 (total dose = 10 g/m2); Vincristine: 2 mg IV by rapid administration on day 0 (for patients with small cell histology).
  Interventions: Drug: Palonosetron - Triple Dose; Drug: Adriamycin; Drug: Ifosfamide chemotherapy (AI); Drug: Zinecard; Drug: Mesna; Drug: Vincristine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Palonosetron - Single Dose — 0.25 mg by vein for 1 dose (day 0).
  Other Names: Aloxi
  Arms: Palonosetron - 1 Dose
Drug: Palonosetron - Triple Dose — 0.25 mg by vein for 3 doses (days 0, 2, 4).
  Other Names: Aloxi
  Arms: Palonosetron - 3 Doses
Drug: Adriamycin — 75 mg/m2 as an IV bolus OR 75 mg/m2 as continuous IV infusion over 72 hours (without zinecard) on Day 0.
  Other Names: Doxorubicin; Doxorubicin Hydrochloride; Adriamycin PFS; Adrimaycin RDF; Rubex
Drug: Ifosfamide chemotherapy (AI) — Ifosfamide: 2.5 g/m2 IV bolus over 3 hours; days 0, 1, 2, 3 (total dose = 10 g/m2). Cycle is 3 weeks, up to 6 cycles.
  Other Names: Ifex
Drug: Zinecard — 750 mg/m2 as an IV bolus.
  Other Names: Dexrazoxane
Drug: Mesna — 500 mg/m2 given simultaneously with ifosfamide day 0; then 1500 mg/m2 over 24 hour for days 0, 1, 2, and 3 (infusion completing on day 4).
  Other Names: mesnex
Drug: Vincristine — 2 mg IV by rapid administration on day 0 (for patients with small cell histology).
  For patients with certain types of sarcoma, vincristine will be given through the catheter by rapid infusion on Day 0 only.
Drug: Dexamethasone — IV piggyback (IVPB) daily for 5 days (12 mg on day 0, and 8 mg on days 1-4) 30 minutes prior to chemotherapy.
  Other Names: Decadron; Dexamethasone acetate

SUMMARY:
The goal of this clinical research study is to compare 2 treatment schedules of Aloxi (palonosetron) in patients with sarcoma who are receiving chemotherapy with adriamycin and ifosfamide. The safety of the drug and schedules will be studied. The effect of palonosetron on patients' quality of life (QOL) will also be studied.

DETAILED DESCRIPTION:
Palonosetron is a drug that is designed to prevent and treat nausea and vomiting that is caused by chemotherapy.

If you are found to be eligible to take part in this study, you will have several blood samples taken (about 3 teaspoons each). Researchers will use the samples to monitor blood counts during chemotherapy and periods of myelosuppression (a condition in which bone marrow activity is decreased). These blood samples will be taken at least 2 times a week, and at certain times, they will be taken once a day. You will be asked to fill out a QOL questionnaire about nausea and vomiting, at least 2 times during Cycle 1 (one cycle lasts 21 days). It will take about 10 minutes to complete the questionnaire.

You will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in one group will receive one dose of palonosetron on Day 0. Participants in the other group will receive 3 doses of palonosetron on Days 0, 2, and 4. Palonosetron will be given to participants in both groups, as an intravenous (IV--through a needle in your vein) infusion over 30 minutes.

You will be asked to keep a study diary during the treatment period. Study personnel will give you the diary and tell you how to complete it. Your side effects (including how severe they are) and medication doses need to be recorded in your diary every day. You will be asked to return your diary at each post-treatment return visit (about every 3 weeks).

While you are on this study, you will receive chemotherapy as part of your standard treatment. All participants will receive at least 2 cycles of adriamycin and ifosfamide chemotherapy (AI). A cycle is 3 weeks long. You may receive up to 6 cycles of adriamycin and ifosfamide. Adriamycin will be given as one large injection through a central venous catheter (plastic tube and needle placed under the collarbone) on Day 0. Ifosfamide will be given over 3 hours every day for 4 days (Days 0-3). Zinecard will be given as one large injection through the catheter on Day 0. Mesna will be given as a 24-hour infusion every day for 4 days through the same catheter (Days 0-3). Zinecard and mesna are given as standard of care. Zinecard is used to protect against heart-related side effects. Mesna is used to protect against bladder-related side effects. For patients with certain types of sarcoma, vincristine will be given through the catheter by rapid infusion on Day 0 only.

You may be treated as an outpatient or an inpatient. You will be asked to return to M. D.Anderson every 3 weeks for evaluation of your disease, by having a chest x-ray, a computerized tomography (CT) scan, a magnetic resonance imaging (MRI) scan, and a physical exam performed. Additional blood samples (about 3 teaspoons) will be taken before each cycle and as often as needed to measure your blood counts and electrolytes (minerals in the body) to monitor any imbalances.

You will be asked to contact the study doctor or nurse about any bad side effects you experience or any medications (over-the-counter or prescription) you take during the treatment period. You will also be asked to notify your other doctors (separate from the study doctors) that you are participating in this research study.

Your treatment will continue for at least 6 cycles, unless your disease gets worse or you experience intolerable side effects. If you experience any intolerable side effects or your disease gets worse while on this study, you may be taken off this study.

Once you stop treatment, you will have what is called an end-of-study visit. During this visit, you will be evaluated for your disease status with CT and MRI scans. You will have your vital signs and weight measured. You will be asked about any medications you have taken since your last visit and any bad side effects that you have experienced. You will also have a final blood draw (about 3 teaspoons) for routine tests.

Your participation in this study should end at about 18 weeks (4 to 5 months).

Once you go off this study, you will have standard follow-up as is required by your doctor.

This is an investigational study. Palonosetron is FDA approved and is commercially available.

Up to 50 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sarcoma which is locally advanced, at high risk for relapse or metastatic for whom treatment with AI is indicated.
* Must be between the ages of 18 and 65 years of age.
* Patients with childbearing potential (defined as not post menopausal for 12 months or no previous surgical sterilization) must use adequate birth control.
* Adequate hematologic (Absolute neutrophil count (ANC)>/= 1500/mm^3, >/= hemoglobin (Hgb, Hb) 10gm/dL, platelet count >/= 150,000/mm^3), renal (serum creatinine </= 1.5 mg/dL), hepatic (serum bilirubin count </= 1.5 * normal and Serum glutamic pyruvic transaminase (SGPT) <3 * normal) functions.
* Karnofsky Performance Status >/= 80.
* Signed informed consent form.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with comorbid condition which renders patients at high risk of treatment complication.
* Patients with symptomatic or untreated metastatic disease to CNS.
* Patients with significant cardiac disease (New York Heart Association (NYHA) Class III or IV), arrhythmia, or recent history of Myocardial infarction (MI) or ischemia.
* Patients with known hypersensitivity to 5-HT3 antagonists.
* Any vomiting or >/= grade 2 nausea in the 24 hours preceding chemotherapy.
* Ongoing vomiting from any organic etiology.
* Radiotherapy within 2 weeks of study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 27, 2006 to March 22, 2011. All recruitment done in medical clinic at UT MD Anderson Cancer Center.
Pre-assignment Details: One participant of the 51 participants recruited withdrew from the trial before assignment to groups and therefore was excluded.
Period: Overall Study
Arm/Group | Palonosetron - 1 Dose | Palonosetron - 3 Doses
Started | 16 | 34
Completed | 16 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palonosetron - 1 Dose | Palonosetron - 3 Doses | Total
Number analyzed (Participants) | 16 | 34 | 50
Age Continuous [Mean (Full Range); unit: years] | 47 [21 to 64] | 52 [22 to 66] | 50 [21 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 15 | 21
  Male | 10 | 19 | 29
Region of Enrollment [Number; unit: participants]
  United States | 16 | 34 | 50

OUTCOME MEASURES:

1. Primary Outcome: Palonosetron Response Rate in the 10 Day Study Cycle
Description: Number of participants with dose of palonosetron who experienced response (no emesis) during acute and delayed time period of the study (10 days) divided by number of participants. Complete response defined as no emesis and no rescue medicines in 10 days from the start of chemotherapy in the first chemotherapy cycle.
Time Frame: 10 days
Measure: Number; unit: percentage of participants
Arm/Group | Palonosetron - 1 Dose | Palonosetron - 3 Doses
Number analyzed (Participants) | 16 | 34
percentage of participants | 31.25 [12.1 to 58.5] | 50 [32.75 to 67.25]

ADVERSE EVENTS:
Time Frame: 3 years and 7 months
Groups:
- Palonosetron: Arm 1: Palonosetron 0.25 mg intravenous (IV) for 1 dose (day 0) and Arm 2: Palonosetron 0.25 mg IV for 3 doses (days 0, 2, 4).
  Dexamethasone: IV piggyback daily for 5 days (12 mg on day 0, and 8 mg on days 1-4) 30 minutes prior to chemotherapy. Chemotherapy treatment regimen: Zinecard: 750 mg/m2 as an IV bolus; Doxorubicin: 75 mg/m2 as an IV bolus OR 75 mg/m2 as continuous IV infusion over 72 hours (without zinecard) on Day 0. Mesna: 500 mg/m2 given simultaneously with ifosfamide day 0; then 1500 mg/m2 over 24 hours for days 0, 1, 2, and 3 (infusion completing on day 4); Ifosfamide: 2.5 g/m2 IV bolus over 3 hours; days 0, 1, 2, 3 (total dose = 10 g/m2); Vincristine: 2 mg IV by rapid administration on day 0 (for patients with small cell histology).
Arm/Group | Palonosetron
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 37/50
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palonosetron (N=50)
Headache (General disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Palpitation (Cardiac disorders) | 1
Fatigue (General disorders) | 2
Constiptation (Gastrointestinal disorders) | 14
Paresthesia (Skin and subcutaneous tissue disorders) | 1
Gastrointestinal Others (Gastrointestinal disorders) | 2 — Altered Taste; Reflux
Weakness (General disorders) | 1
Skin Changes (Skin and subcutaneous tissue disorders) | 1
Indigestion (Gastrointestinal disorders) | 1
Hiccups (General disorders) | 1
Sweat (General disorders) | 1
Anorexia (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes